CLINICAL TRIAL: NCT06946797
Title: A Phase 2, Open-label, Randomized Trial to Evaluate Two Dosing Regimens of Subcutaneous Formulation of Nivolumab in Combination With Intravenous Ipilimumab and Chemotherapy in Participants With Previously Untreated Metastatic or Recurrent NSCLC
Brief Title: A Study to Evaluate Two Dosing Regimens of Subcutaneous Nivolumab in Combination With Intravenous Ipilimumab and Chemotherapy in Participants With Previously Untreated Metastatic or Recurrent Non-Small Cell Lung Cancer (NSCLC)
Acronym: CheckMate-1533
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-1533
Record Dates: First submitted 2025-04-25; First posted 2025-04-27 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Nivolumab; Ipilimumab; Checkmate-1533; CA2091533; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Ipilimumab; Carboplatin; Paclitaxel; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Pemetrexed; Drug: Cisplatin
- Arm B (Experimental)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Nivolumab — Specified dose on specified days
  Other Names: BMS-986298
Drug: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy
Drug: Carboplatin — Specified dose on specified days
Drug: Paclitaxel — Specified dose on specified days
Drug: Pemetrexed — Specified dose on specified days
Drug: Cisplatin — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate two dosing regimens of subcutaneous Nivolumab in combination with intravenous Ipilimumab and chemotherapy in participants with previously untreated metastatic or recurrent Non-Small Cell Lung Cancer (NSCLC)

ELIGIBILITY:
Inclusion Criteria

* Participants must have histologically confirmed stage IV or recurrent non-small cell lung cancer (NSCLC) (as defined by the 9th edition of the IASLC Lung Cancer Staging Guidelines) of squamous or non-squamous histology.
* Participants must have no prior systemic anti-cancer treatment (including EGFR, ALK, ROS-1, BRAF, RET, and NTRK inhibitors) given as primary therapy for advanced or metastatic disease.
* Participants with prior definitive chemoradiation for locally advanced disease is permitted as long as the last administration of chemotherapy or radiotherapy (whichever was given last) occurred at least 6 months prior to randomization. Participants with locally advanced disease with recurrence after chemoradiation therapy (stage III disease, specifically refers to patients with no curative options) are eligible to enroll.
* Participants with prior adjuvant or neoadjuvant chemotherapy for early-stage lung cancer are permitted if completed at least 6 months prior to randomization.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1 at screening and confirmed prior to randomization.
* Participants must have measurable disease by CT or MRI per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria with radiographic tumor assessment performed within 28 days of randomization.

Exclusion Criteria

* Participants must not have any prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Participants must not have any known driver mutations with available targeted therapy (including but not limited to EGFR mutations, ALK translocations, ROS-1 translocations and known BRAFV600E, that are sensitive to available targeted inhibitor therapy; participants with a known activating RET mutations and NTRK fusion gene alterations).
* Participants must not have any untreated central nervous system (CNS) metastases
* Participants must not have leptomeningeal metastases (carcinomatous meningitis).
* Participants must not have any active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Participants with previous malignancies (except non-melanoma skin cancers, and in situ cancers such as the following: bladder, gastric, colon, cervical/dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to randomization and no additional therapy is required or anticipated to be required during the study period.
* Participants must not have a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) within 14 days or other immunosuppressive medications within 30 days of randomization. Inhaled or topical steroids, and adrenal replacement steroid > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Participants must not have any history of interstitial lung disease or pneumonitis that required oral or IV glucocorticoids to assist with management.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2027-02-05 (Estimated); Study Completion 2028-10-25 (Estimated)

PRIMARY OUTCOMES:
Maximum observed serum concentration (Cmax) of subcutaneous Nivolumab in serum | Up to 3 weeks
Time to peak concentration (Tmax) of subcutaneous Nivolumab in serum | Up to 3 weeks
Area under the concentration-time curve within a dosing interval (AUC(TAU)) of subcutaneous Nivolumab in serum | Up to 3 weeks
Concentration at the end of a dosing interval (Ctau) of subcutaneous Nivolumab in serum | Up to 3 weeks
Trough observed concentration (Ctrough) of subcutaneous Nivolumab | At Cycle 7 Day 1 (Week 18)

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to approximately 2.5 years
Number of participants with serious adverse events (SAEs) | Up to approximately 2.5 years
Number of participants with drug related AEs | Up to approximately 2.5 years
Number of participants with Immune Mediated Adverse Events (IMAEs) | Up to approximately 2.5 years
Number of participants with AEs leading to discontinuation | Up to approximately 2.5 years
Number of deaths | Up to approximately 2.5 years
Number of participants with anti-nivolumab antibodies | Up to approximately 2.5 years
Number of participants with anti-ipilimumab antibodies | Up to approximately 2.5 years
Number of participants with neutralizing antibodies | Up to approximately 2.5 years
Cmax of intravenous Ipilimumab in serum | Up to 6 weeks
Tmax of intravenous Ipilimumab in serum | Up to 6 weeks
AUC(TAU) of intravenous Ipilimumab in serum | Up to 6 weeks
Ctau of intravenous Ipilimumab in serum | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (50):
- United States (9):
  - Alaska Oncology and Hematology, Anchorage, Alaska
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Local Institution - 0088, Newport Beach, California
  - Local Institution - 0063, Boise, Idaho
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Local Institution - 0064, Post Falls, Idaho
  - Local Institution - 0047, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
- Brazil (5):
  - Local Institution - 0041, Brasília, Federal District
  - Local Institution - 0043, Belo Horizonte, Minas Gerais
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Icesp - Instituto Do Câncer Do Estado de São Paulo, São Paulo
- Chile (3):
  - Local Institution - 0068, Antofagasta, AN
  - Local Institution - 0069, Viña del Mar, Región de Valparaíso
  - Local Institution - 0067, Santiago, Santiago Metropolitan
- France (3):
  - Centre Georges François Leclerc, Dijon, Côte-d'Or
  - Hôpital Foch, Suresnes, Hauts-de-Seine
  - Groupe hospitalier Paris saint Joseph, Paris, Île-de-France Region
- Greece (4):
  - Thoracic General Hospital of Athens "I Sotiria", Athens, Attikí
  - Local Institution - 0013, Chaïdári, Attikí
  - Local Institution - 0011, Thessaloniki, Kentrikí Makedonía
  - University General Hospital of Larissa, Larissa, Thessalía
- Italy (5):
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola, Emilia-Romagna
  - P.O. "S. Maria della Misericordia" Azienda Sanitaria Universitaria Friuli Centrale, Udine, Friuli Venezia Giulia
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo, Lombardy
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliero Universitaria Maggiore della Carità, Novara
- Mexico (5):
  - Local Institution - 0025, Guadalajara, Jalisco
  - Local Institution - 0058, Monterrey, Nuevo León
  - Local Institution - 0027, Mérida, Yucatán
  - Local Institution - 0024, México
  - Local Institution - 0022, Puebla City
- Poland (3):
  - Local Institution - 0081, Warsaw, Masovian Voivodeship
  - Szpital Specjalistyczny w Prabutach Spolka z o.o., Prabuty, Pomeranian Voivodeship
  - Instytut Centrum Zdrowia Matki Polki, Lodz, Łódź Voivodeship
- Romania (6):
  - Institutul Oncologic Bucuresti, Bucharest, București
  - SC Radiotherapy Center Cluj SRL, Florești, Cluj
  - Centrul de Oncologie "Sfântul Nectarie", Craiova, Dolj
  - Centrul de Diagnostic si Tratament Provita, Bucharest
  - Institutul Oncologic Cluj, Cluj-Napoca
  - Institutul Regional de Oncologie, Iași
- South Africa (4):
  - Local Institution - 0066, Pretoria, Gauteng
  - Local Institution - 0031, Soweto, Gauteng
  - Local Institution - 0009, Sandton, GP
  - Cancercare Rondebosch Oncology, Rondebosch, Western Cape
- Turkey (Türkiye) (3):
  - Local Institution - 0070, Adana
  - Local Institution - 0072, Ankara
  - Local Institution - 0071, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06946797.html